CLINICAL TRIAL: NCT07374991
Title: Clinical and Molecular Effects of N-Acetylcysteine Treatment in COVID-19-Related Acute Respiratory Distress Syndrome: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Clinical and Molecular Effects of N-Acetylcysteine Treatment in COVID-19-Related Acute Respiratory Distress Syndrome
Acronym: A Prospective
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Gülseren, prof, University of Gaziantep
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: TF.20.26
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: COVID-19-Associated Acute Respiratory Distress Syndrome (ARDS)

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Double-blind (participant, care provider, investigator, outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine (NAC) Group (Experimental): Participants received intravenous N-acetylcysteine (150 mg/kg on day 1, followed by 50 mg/kg/day on days 2 and 3) in addition to standard of care.
  Interventions: Diagnostic Test: N-Acetylcysteine (NAC)
- Plasebo (Placebo Comparator): Participants received intravenous 0.9% sodium chloride (placebo) administered at the same volume and duration as the intervention group, in addition to standard of care.
  Interventions: Diagnostic Test: N-Acetylcysteine (NAC)

INTERVENTIONS:
Diagnostic Test: N-Acetylcysteine (NAC) — Intravenous N-acetylcysteine administered at 150 mg/kg on day 1 followed by 50 mg/kg/day on days 2 and 3, in addition to standard of care.
  Other Names: NAC

SUMMARY:
Prospective, randomized, double-blind, placebo-controlled clinical trial evaluating the clinical and molecular effects of intravenous N-acetylcysteine (NAC) in patients with COVID-19-associated acute respiratory distress syndrome (ARDS) treated in the intensive care unit. The study assessed inflammatory and thromboinflammatory biomarkers, hypoxia-related gene expression (HIF-1α, ACE2, CD147), and clinical outcomes including mortality and length of ICU stay.

DETAILED DESCRIPTION:
This single-center, prospective, randomized, double-blind, placebo-controlled clinical trial was conducted in adult patients with PCR-confirmed COVID-19 and acute respiratory distress syndrome (ARDS) admitted to the intensive care unit. Eligible patients were randomly assigned in a 1:1 ratio to receive intravenous N-acetylcysteine (NAC) or placebo in addition to standard care. NAC was administered at a dose of 150 mg/kg on day 1 followed by 50 mg/kg/day on days 2 and 3.

The primary objectives were to evaluate the effects of NAC on inflammatory and thromboinflammatory biomarkers and hypoxia-related molecular pathways. Biochemical parameters including C-reactive protein, D-dimer, ferritin, zinc levels, and PaO₂/FiO₂ ratio were measured at ICU admission and on day 4. Gene expression levels of HIF-1α, ACE2, and CD147 were analyzed in peripheral blood using RT-qPCR.

Secondary objectives included assessment of clinical outcomes such as mortality, length of intensive care unit stay, and need for mechanical ventilation. The study was approved by the institutional ethics committee, and written informed consent was obtained from patients or their legal representatives.

ELIGIBILITY:
Inclusion Criteria:Age ≥18 years

PCR-confirmed SARS-CoV-2 infection

Diagnosis of acute respiratory distress syndrome (ARDS) according to the Berlin criteria

Admission to the intensive care unit

Written informed consent obtained from the patient or legal representative -

Exclusion Criteria:Expected mortality within 48 hours of ICU admission

Prior chronic oxygen therapy

Previous COVID-19 treatment initiated at another center

Pregnancy or breastfeeding

Use of antioxidant or anti-inflammatory drugs within 30 days prior to enrollment

Known hypersensitivity to N-acetylcysteine

Use of medications affecting glutathione metabolism

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory and thromboinflammatory biomarkers | Baseline (ICU admission) to Day 4
  Change in C-reactive protein (CRP) and D-dimer levels from baseline (ICU admission) to day 4 of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep üniversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No